CLINICAL TRIAL: NCT00168948
Title: Intermittent Treatment With Sulfadoxine-Pyrimethamine for Malaria Control in Children: A Randomised, Double Blind, and Placebo-Controlled Clinical Trial
Brief Title: Intermittent Antimalaria Treatment With SP in African Children
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Deutscher Akademischer Austausch Dienst (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 01KA0202-T; 01KA0202
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2005-11-02 (Estimated); Status verified 2003-02

CONDITIONS: Malaria; Anemia
Keywords: Intermittent preventive treatment; IPTi; Malaria control; Ghana
MeSH Terms: conditions — Malaria; Anemia | interventions — Pyrimethamine

INTERVENTIONS:
Drug: Sulfadoxin (12.5) Pyrimethamine (250 mg)

SUMMARY:
- intermittent preventive treatment with SP in children to evaluate efficacy and safety of this drug combination in children in northern Ghana

DETAILED DESCRIPTION:
* Sulfadoxine and pyrimethamine have long been used for malaria prevention and treatment. In this study, following suggestions of WHO, these drugs are used for intermittent treatment.
* It will be tested if this approach reduces the number of malaria attacks and ameliorates the severity of the disease
* It will also be determined if anemia due to malaria, which is prevalent in northern Ghana, may be reduced
* Moreover, the interaction between red cell polymorphisms such as HbS, HbC, alpha-thalassemia and glucose-6-phosphate dehydrogenase deficiency and SP will be examined

ELIGIBILITY:
Inclusion Criteria:

* informed consent by parents or guardian
* no concomitant serious disease
* age >2 months

Exclusion Criteria:

* serious allergy or hypersensitivity to sulfonamides or pyrimethamine
* no severe hepatic or renal dysfunction
* serious breach of study protocol

Ages: 2 Months to 4 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1200
Dates: Start 2003-03; Study Completion 2005-08

PRIMARY OUTCOMES:
Efficacy and safety of IPTi with SP
Impact of IPTi on incidence on malaria attacks
Impact of IPTi on anemia

SECONDARY OUTCOMES:
Interaction between erythrocyte polymorphisms and SP
Influence on parasite multiplicity
Impact on child development

CONTACTS AND LOCATIONS:
Overall Officials: Frank Mockenhaupt, PhD, Study Director — Charite University-Medicine, Berlin, Germany

REFERENCES:
- [Background] Schellenberg D, Menendez C, Kahigwa E, Aponte J, Vidal J, Tanner M, Mshinda H, Alonso P. Intermittent treatment for malaria and anaemia control at time of routine vaccinations in Tanzanian infants: a randomised, placebo-controlled trial. Lancet. 2001 May 12;357(9267):1471-7. doi: 10.1016/S0140-6736(00)04643-2. PMID 11377597
- [Background] Menendez C, Kahigwa E, Hirt R, Vounatsou P, Aponte JJ, Font F, Acosta CJ, Schellenberg DM, Galindo CM, Kimario J, Urassa H, Brabin B, Smith TA, Kitua AY, Tanner M, Alonso PL. Randomised placebo-controlled trial of iron supplementation and malaria chemoprophylaxis for prevention of severe anaemia and malaria in Tanzanian infants. Lancet. 1997 Sep 20;350(9081):844-50. doi: 10.1016/S0140-6736(97)04229-3. PMID 9310602
- [Background] Massaga JJ, Kitua AY, Lemnge MM, Akida JA, Malle LN, Ronn AM, Theander TG, Bygbjerg IC. Effect of intermittent treatment with amodiaquine on anaemia and malarial fevers in infants in Tanzania: a randomised placebo-controlled trial. Lancet. 2003 May 31;361(9372):1853-60. doi: 10.1016/s0140-6736(03)13504-0. PMID 12788572